CLINICAL TRIAL: NCT02393105
Title: The Sense of Hope Alleviates Fatigue in Breast Cancer Survivors
Brief Title: Sense of Hope Alleviates Fatigue in Breast Cancer Survivors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201411051RINB
Record Dates: First submitted 2015-01-06; First posted 2015-03-19 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Carcinoma of Male Breast
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms, Male; Breast Neoplasms

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Breast cancer survivor: Females finished primary breast cancer treatment including surgical operation, radiation therapy and chemotherapy.

SUMMARY:
This study explores the relationship between the sense of hope and fatigue in breast cancer survivors and provides a reference for future planning improvements for breast cancer survivors experiencing fatigue.

DETAILED DESCRIPTION:
Breast cancer is an important and escalating issue for females all over the world. Due to the improvement of medical and technological progress, the survival rate of breast cancer patient increases every year. Breast cancer survivors, after the discomforting distress from cancer treatment, will go through treatment-derived physical distress and worry about relapse. As a result the fatigue in breast cancer survivors has not been reduced after primary treatment. Feeling fatigue in a long term will bring mental illness problems ,decrease the quality of life and weaken the will to survive. A sense of hope in the face of fatigue may serve as an important driving force and enhance the survivors' will to survive. This study explores the relationship between the sense of hope and fatigue in breast cancer survivors and provides a reference for future planning improvements for breast cancer survivors experiencing fatigue.

A cross-sectional study design is adopted for this study. The study expects to collect 200 questionnaires from breast cancer survivors through medical centers treating breast cancer and breast cancer patients communities. The questionnaire includes (a) the basic demographic information (b) disease history (c) social support scale; (d) short version multiaxial fatigue syndrome scale; (e) Hearst hope scale.

Answered questionnaires will be input to spreadsheets for further statistical analysis using SPSS 19.0 statistical software packages.

ELIGIBILITY:
Inclusion criteria:

1. diagnosed as a breast cancer patient
2. complete operation,chemotherapy and radiation therapy
3. understand the treatment and condition by herself
4. conscious clear who can speaking Mandarin or: Taiwanese
5. after consenting , the participant agree to participate orally or write down in the consent form

Exclusion criteria:

1. Can not speaking Mandarin or Taiwanese
2. Psychotic or Understanding barriers
3. refuse verbally or write the Consent Form

Ages: 20 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: breast cancer survivors,complete chemotherapy and radiotherapy
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Multidimensional Fatigue Symptom Inventory-Short Form | Baseline measured after the completion of breast cancer surgery, radiation therapy and chemotherapy
  A 30-item self-report questionnaire designed to assess the severity, frequency, and daily pattern of fatigue as well as its perceived interference with quality of life.

SECONDARY OUTCOMES:
Herth Hope Index | Baseline measured after the completion of breast cancer surgery, radiation therapy and chemotherapy
  A 12-item self-report questionnaire containing three dimensions: temporality and future, positive readiness and expectancy, and interconnectedness. Tested on family caregivers of terminally ill people and terminally ill persons as well as in community and hospital patients and family members. (Herth, 1990)
The Inventory of Socially Supportive Behaviors | Baseline measured after the completion of breast cancer surgery, radiation therapy and chemotherapy
  A 40-item self-report questionnaire designed to assess how often individuals received various forms of assistance during the preceding month, such as directive guidance (e.g., offering advice), nondirective support (e.g., listening and reflecting), positive social exchange (e.g., expressing confidence and encouragement), and tangible assistance (e.g., providing materials or services). (Barrera, Sandler, & Ramsay, 1981).

CONTACTS AND LOCATIONS:
Overall Officials: ChunaNG Pei-Hsuan, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Alexander S, Minton O, Andrews P, Stone P. A comparison of the characteristics of disease-free breast cancer survivors with or without cancer-related fatigue syndrome. Eur J Cancer. 2009 Feb;45(3):384-92. doi: 10.1016/j.ejca.2008.09.010. Epub 2008 Oct 30. PMID 18977131
- [Background] Berger AM, Gerber LH, Mayer DK. Cancer-related fatigue: implications for breast cancer survivors. Cancer. 2012 Apr 15;118(8 Suppl):2261-9. doi: 10.1002/cncr.27475. PMID 22488700
- [Background] Brady MJ, Peterman AH, Fitchett G, Mo M, Cella D. A case for including spirituality in quality of life measurement in oncology. Psychooncology. 1999 Sep-Oct;8(5):417-28. doi: 10.1002/(sici)1099-1611(199909/10)8:53.0.co;2-4. PMID 10559801
- [Background] Dizon DS. Quality of life after breast cancer: survivorship and sexuality. Breast J. 2009 Sep-Oct;15(5):500-4. doi: 10.1111/j.1524-4741.2009.00766.x. Epub 2009 Jul 14. PMID 19614908
- [Background] Gielissen MF, Wiborg JF, Verhagen CA, Knoop H, Bleijenberg G. Examining the role of physical activity in reducing postcancer fatigue. Support Care Cancer. 2012 Jul;20(7):1441-7. doi: 10.1007/s00520-011-1227-4. Epub 2011 Jul 21. PMID 21773676
- [Background] Goldstein D, Bennett BK, Webber K, Boyle F, de Souza PL, Wilcken NR, Scott EM, Toppler R, Murie P, O'Malley L, McCourt J, Friedlander M, Hickie IB, Lloyd AR. Cancer-related fatigue in women with breast cancer: outcomes of a 5-year prospective cohort study. J Clin Oncol. 2012 May 20;30(15):1805-12. doi: 10.1200/JCO.2011.34.6148. Epub 2012 Apr 16. PMID 22508807
- [Background] Hoffman AJ, von Eye A, Gift AG, Given BA, Given CW, Rothert M. Testing a theoretical model of perceived self-efficacy for cancer-related fatigue self-management and optimal physical functional status. Nurs Res. 2009 Jan-Feb;58(1):32-41. doi: 10.1097/NNR.0b013e3181903d7b. PMID 19092553
- [Background] Howard-Anderson J, Ganz PA, Bower JE, Stanton AL. Quality of life, fertility concerns, and behavioral health outcomes in younger breast cancer survivors: a systematic review. J Natl Cancer Inst. 2012 Mar 7;104(5):386-405. doi: 10.1093/jnci/djr541. Epub 2012 Jan 23. PMID 22271773
- [Background] Koch L, Jansen L, Herrmann A, Stegmaier C, Holleczek B, Singer S, Brenner H, Arndt V. Quality of life in long-term breast cancer survivors - a 10-year longitudinal population-based study. Acta Oncol. 2013 Aug;52(6):1119-28. doi: 10.3109/0284186X.2013.774461. Epub 2013 Mar 20. PMID 23514583
- [Background] Mattioli JL, Repinski R, Chappy SL. The meaning of hope and social support in patients receiving chemotherapy. Oncol Nurs Forum. 2008 Sep;35(5):822-9. doi: 10.1188/08.ONF.822-829. PMID 18765329
- [Background] Olson K. A new way of thinking about fatigue: a reconceptualization. Oncol Nurs Forum. 2007 Jan;34(1):93-9. doi: 10.1188/07.ONF.93-99. PMID 17562637
- [Background] Piper BF, Cella D. Cancer-related fatigue: definitions and clinical subtypes. J Natl Compr Canc Netw. 2010 Aug;8(8):958-66. doi: 10.6004/jnccn.2010.0070. PMID 20870639
- [Background] Ribi K, Bernhard J, Rufibach K, Thurlimann B, von Moos R, Ruhstaller T, Glaus A, Bohme C. Endocrine symptom assessment in women with breast cancer: what a simple "yes" means. Support Care Cancer. 2007 Dec;15(12):1349-56. doi: 10.1007/s00520-007-0258-3. Epub 2007 May 26. PMID 17530302
- [Background] Rustoen T, Cooper BA, Miaskowski C. The importance of hope as a mediator of psychological distress and life satisfaction in a community sample of cancer patients. Cancer Nurs. 2010 Jul-Aug;33(4):258-67. doi: 10.1097/NCC.0b013e3181d6fb61. PMID 20467303
- [Background] Trudel-Fitzgerald C, Savard J, Ivers H. Evolution of cancer-related symptoms over an 18-month period. J Pain Symptom Manage. 2013 Jun;45(6):1007-18. doi: 10.1016/j.jpainsymman.2012.06.009. Epub 2012 Sep 24. PMID 23017613